CLINICAL TRIAL: NCT05735652
Title: An Observational Study to Evaluate the Safety and Effectiveness of Radiotherapy for Localized T1-T2 Prostate Cancer in China After Injection of SpaceOAR Hydrogel
Brief Title: An Observational Study of Radiotherapy After Injection of SpaceOAR Hydrogel
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: U0745
Record Dates: First submitted 2022-08-22; First posted 2023-02-21 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with localized T1-T2 prostate cancer in China who were injected with SpaceOAR Hydrogel: This observational study aims to evaluate the safety and effectiveness of radiotherapy for subjects with localized T1-T2 prostate cancer in China who were injected with SpaceOAR Hydrogel, via collecting clinical data related to radiotherapy.
  Interventions: Device: SpaceOAR Hydrogel

INTERVENTIONS:
Device: SpaceOAR Hydrogel — The SpaceOAR System is an in-situ formed absorbable hydrogel that is administered transperineally (with transrectal ultrasound guidance) between the prostate and rectum

SUMMARY:
This observational study aims to evaluate the safety and effectiveness of radiotherapy for subjects with localized T1-T2 prostate cancer in China who were injected with SpaceOAR Hydrogel, via collecting clinical data related to radiotherapy.

DETAILED DESCRIPTION:
This study protocol is for the second part of SpaceOAR real world study in which long term follow-up visits will be performed (up to 1 year) outside Boao Medical Tourism Pilot Zone. The SpaceOAR real world study is a retrospective and prospective, single arm, observational study (Ptotocol of SpaceOAR RWS Windchill#: 92743236). Subjects with localized T1-T2 prostate cancer who have already been injected with the SpaceOAR and have received radiotherapy or will receive radiotherapy will be enrolled, and clinical data related to radiotherapy will be collected. For subjects who have already completed radiotherapy before study kick-off, clinical data will be collected retrospectively, such as data related to radiotherapy, AE (if any) and MRI (if any). Follow up vist will be completed if applicable. For subjects who receive therapy after study kick-off, follow up visits at 2 weeks, 6weeks, 3 months and 10 months after radiotherapy will be scheduled to assess bowel, urinary and sexual function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have provided the written informed consent, are willing to participate in clinical data collection and willing to comply with study procedure. (for subjects enrolled prospectively)
* Subjects must have been pathologically confirmed prostate cancer with clinical stage T1-T2, and have been treated with Space OAR Hydrogel, and have received or will receive radiotherapy.

Exclusion Criteria:

* All subjects have received radiotherapy or will receive radiotherapy, who have injected with SpaceOAR hydrogel in Boao Medical Pilot Zone.
* There is no specific exclusion criteria unless the patients refuse to sign the informed consent.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: During screening, patients who have received or will receive radiotherapy will be identified.
  These who have been injected with SpaceOAR hydrogel will be enrolled. For patients who have already received radiotherapy, the clinical data can be collected retrospectively, and informed consent will be performed (If follow up visits can be conducted prospectively). For patients who will receive radiotherapy, informed consent will be gained.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nianzeng Xing, Doctor, Principal Investigator — Hospital Executive
Locations (1):
- Shanxi Cancer Hospital, Taiyuan, Shanxi, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects for this study are patients with localized prostate cancer enrolled in the SpaceOAR Hainan Real World Study (U0720) who have been treated with SpaceOAR hydrogel at a hospital in the Boao Lecheng Medical Pilot Area in Hainan and have received or will receive radiation therapy at the study center.
Groups:
- Observational Study of 14 Cases, Single Arm: This observational study single arm aims to evaluate the safety and effectiveness of radiotherapy for subjects with localized T1-T2 prostate cancer in China who were injected with SpaceOARHydrogel, via collecting clinical data related to radiotherapy.
Period: Overall Study
Arm/Group | Observational Study of 14 Cases, Single Arm
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: For subjects who have already completed radiotherapy before study kick-off, clinical data will be collected retrospectively, such as data related to radiotherapy, AE (if any) and MRI (if any), and follow up will be performed, if applicable.
  For subjects who receive therapy after study kick-off, radiotherapy relevant clinical data will be collected, and follow up visits after radiotherapy will be scheduled to assess urinary, bowel, sexual functions and AE.
Groups:
- Single Arm Obsevational Study Total 14 Cases: This observational single arm study aims to evaluate the safety and effectiveness of radiotherapy for subjects with localized T1-T2 prostate cancer in China who were injected with SpaceOAR Hydrogel, via collecting clinical data related to radiotherapy.
  SpaceOAR Hydrogel: The SpaceOAR System is an in-situ formed absorbable hydrogel that is administered transperineally (with transrectal ultrasound guidance) between the prostate and rectum.
Arm/Group | Single Arm Obsevational Study Total 14 Cases
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (7.9)
Sex/Gender, Customized [Count of Participants; unit: Participants] — The study indication was prostate cancer, so all enrolled patients were male
  Participants
    Count of Participants: Male | 14
    Count of Participants: Female | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change of Dose Rectum Volume Receiving Radiation Between Radiotherapy Plannings Pre and Post SpaceOAR Hydrogel Injection.
Description: Change of dose rectum volume receiving radiation,which is measured by Dose-volume histogram in radiotherapy planning pre and post SpaceOAR hydrogel injection radiotherpy planning is made based on CT simulation scans.
Time Frame: Post injection gel surgery 1-10 days
Population: Potential subjects for this study are patients with localized prostate cancer enrolled in the SpaceOAR Hainan Real World Study (U0720) who have been treated with SpaceOAR hydrogel at a hospital in the Boao Licheng Medical Pilot Area in Hainan and have received or will receive radiation therapy at the study center.
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Subjects With Localized T1-T2 Prostate Cancer in China Who Were Injected With SpaceOAR Hydrogel
Number analyzed (Participants) | 14
cc
  Rectum wall V37Gy (cc) | 2.4 (2.8)
  Rectum wall V46Gy (cc) | 2.7 (2.5)

2. Secondary Outcome: Urinary, Bowel and Sexual Function Assessment Score
Description: Descrpition of change of urinary, bowel and Sexual function assessment score, which are measured by Expanded Prostate cancer Index Composite (EPIC)-26. EPIC-26 is short form version to measure health related quality of life among men with prostate cancer, which contains 26 item and 5 domains : Urinary Incontinence, Urinary irritative/Obstructive, Bowel, Sexual, and Hormonal. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly from 0 score to 100 scores, with higher scores representing better.
Time Frame: After the completion of radiotherapy, the month 3 Expanded Prostate Cancer Index Composite (EPIC)-26 score was compared to the baseline EPIC-26 score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Observational Study of 14 Cases, Single Arm
Number analyzed (Participants) | 14
score on a scale
  Bowel function | 99.4 (1.5)
  Urinary Incontinence | 92.9 (12.7)
  Urinary rritative /Obstructive | 96.0 (5.3)
  Sexual | 31 (16.1)

3. Secondary Outcome: Quality of Life Was Measured by EQ-5D-5L Scale（the Five-level Version of the EuroQol 5-Dimension Scale)
Description: Frequencies and proportions of responses in five dimension (Mobility, Anxiety/Depression, Pain/Discomfort, Usual Activities and Self-Care) and different levels will be tabulated, which was measured by EQ-5D-5L scale（the five-level version of the EuroQol 5-Dimension scale).The minimum value and maximum value of EQ VAS (EQ visual analogue scale) are from 0 score to100 scores, which a higher value means a beter outcome.
Time Frame: After the completion of radiotherapy, the month 3 EQ-5D-5L scale（the five-level version of the EuroQol 5-Dimension scale) score was compared to the baseline EQ-5D-5L scale score.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Obsevational Study Total 14 Cases
Number analyzed (Participants) | 14
score on a scale | 1.0 (0.0)

4. Secondary Outcome: The Distance Between Prostate and Rectum
Description: The distance between the posterior prostatic capsule and anterior rectal wall is measured on the axial image slice closest to halfway between apex and base, from posterior edge of prostate to inner rectal wall via MRI.
Time Frame: After the completion of radiotherapy, the weeks 6 the distance between prostate and rectum measured by MRI was compared to the baseline the distance between prostate and rectum measured by MRI.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Subjects With Localized T1-T2 Prostate Cancer in China Who Were Injected With SpaceOAR Hydrogel
Number analyzed (Participants) | 14
mm | 5.4 (3.8)

5. Secondary Outcome: the Distance Between the Prostate and Rectum
Description: The presence of SpaceOAR hydrogel between prostate and rectum is evaluated by MRI via distance indirectly.
Time Frame: After the completion of radiotherapy, the month 10 the distance between prostate and rectum measured by MRI was compared to the baseline the distance between prostate and rectum measured by MRI.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Subjects With Localized T1-T2 Prostate Cancer in China Who Were Injected With SpaceOAR Hydrogel
Number analyzed (Participants) | 14
mm | 2.0 (1.2)

6. Secondary Outcome: Adverse Event Related to SpaceOAR Hydrogel (Safety)
Description: The relationship of AE /ADE/SAE/SADE/UADEs will be assessed by investigators.
Time Frame: Through the entire study phase until 10 months after the completion of radiotherapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Localized T1-T2 Prostate Cancer in China Who Were Injected With SpaceOAR Hydrogel
Number analyzed (Participants) | 14
Participants | 0

ADVERSE EVENTS:
Time Frame: Through the entire study phase until 10 months after the completion of radiotherapy.
Arm/Group | Subjects With Localized T1-T2 Prostate Cancer in China Who Were Injected With SpaceOAR Hydrogel
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Localized T1-T2 Prostate Cancer in China Who Were Injected With SpaceOAR Hydrogel (N=14)
compression fracture of the lumbo2 vertebrae (Surgical and medical procedures) | 1 (1) — No metastasis was assessed by the investigators, independent of hydrogel and radiation therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Localized T1-T2 Prostate Cancer in China Who Were Injected With SpaceOAR Hydrogel (N=14)
Coronavirus 2019 (COVID-19) (Infections and infestations) | 4 (4) — Coronavirus 2019 (COVID-19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT05735652/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT05735652/SAP_001.pdf